CLINICAL TRIAL: NCT00890279
Title: Phase II Study for the Second-Line Treatment of Hypertension in Patients With Autosomal Dominant Polycystic Kidney Disease; ACEI vs. CCB
Brief Title: Efficacy and Safety Study of Second-Line Treatment for Hypertension With Autosomal Dominant Polycystic Kidney Disease(ADPKD)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ministry of Health, Labour and Welfare, Japan (Other Government)
Responsible Party: Shigeo Horie, M.D./Chairman of the Department of Urology at Teikyo University, Teikyo University, School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ADPKDhypertension
Record Dates: First submitted 2009-04-28; First posted 2009-04-29 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-12

CONDITIONS: Kidney, Polycystic, Autosomal Dominant
Keywords: Autosomal Dominant Polycystic Kidney Disease; Hypertension; Angiotensin-II Receptor Blocker; Calcium Channel Blocker; Angiotensin converting enzyme inhibitor; Kidney Volume; eGFR
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant; Hypertension | interventions — cilnidipine; imidapril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cilnidipine (Experimental): The patients whose blood pressure is not controlled under 120/80 with ARB alone are randomized into group A or B. In group A, blood pressure is controlled by Candesartan plus Cilnidipine.
  Interventions: Drug: Cilnidipine
- Imidapril (Active Comparator): The patients whose blood pressure is not controlled under 120/80 with ARB alone are randomized into group A or B. In group B, blood pressure is controlled by Candesartan plus Imidapril.
  Interventions: Drug: Imidapril

INTERVENTIONS:
Drug: Cilnidipine — Cilnidipine up to 20 mg
  Other Names: ATELEC
  Arms: Cilnidipine
Drug: Imidapril — Imidapril up to 10 mg per day
  Other Names: TANATRIL
  Arms: Imidapril

SUMMARY:
This phase II study examines the safety and efficacy of combination therapy for hypertension in patients with autosomal dominant polycystic kidney disease (ADPKD). This study examines the safety and efficacy of combination therapy by imidapril (ACEI) or cilnidipine (CCB) in ADPKD patients whose blood pressure is not controlled under 120/80 mmHg by candesartan (ARB) alone.

DETAILED DESCRIPTION:
Maximum dosage of candesartan is 8 mg/day. Dosage of imidapril is in the range of 2.5-10 mg/day. Dosage of cilnidipine is in the range of 5-20mg/day.

ELIGIBILITY:
Inclusion Criteria:

* ADPKD patients
* Blood pressure measured at out-patient setting is above 120/80 mmHg
* Age between 20 and 60 years old
* eGFR more than 30 ml/min/1.73m2
* Patients give informed consent

Exclusion Criteria:

* Patients with severe cardiovascular and hepatic disorders
* Patients with complications of central nervous vascular disorders
* Women who are breast feeding and females of childbearing potential who are not using acceptable contraceptive methods
* Patients currently engaging in other experimental protocol
* Patients with intracranial aneurysma
* Patients who must use diuretics
* Allergic patients to Candesartan or Cilnidipine
* Patients whose hypertension is not controlled by medication of this protocol

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-06 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
eGFR | every 6 months

SECONDARY OUTCOMES:
Kidney Volume measured by MRI | every 3 months to every 2 years
Serum creatinine level | every 3 months to every 2 years
Induction of hemodialysis, cardiovascular events and central nervous vascular events | every 3 months to every 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Shigeo Horie, MD, Study Chair — Teikyo University
Locations (9):
- Japan (9):
  - Department of Urology, National Hospital Organaization Chiba-East Hospital, Chiba, Chiba
  - Department of Medicine II, Hokkaido Univserity School of Medicine, Sapporo, Hokkaido
  - Toranomon Hospital Kajigaya, Kidney center, Kawasaki, Kanagawa
  - Division of Clinical Nephrology and Rheumatology, Niigata University Graduate School of Medical and Dental Sciences, Niigata, Niigata
  - Department of Medicine II, Nippon Medical School, Bunkyo-ku, Tokyo
  - Department of Urology, Teikyo University School of Medicine, Itabashi-ku, Tokyo
  - Toranomon Hospital, Kidney center, Minato-ku, Tokyo
  - Division of Kidney and Hypertension, Department of Internal Medicine, Jikei University School of Medicine, Minato-ku, Tokyo
  - Department of Urology, Kyorin University School of Medicine, Mitaka, Tokyo